CLINICAL TRIAL: NCT03526406
Title: Investigation of the Acute and Chronic Cognitive and Mood Effects of CP9700 in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Polyphenolics, Inc. (Industry)
Responsible Party: Principal Investigator, Prof Claire Williams, Chair of Neuroscience, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RDG-003
Record Dates: First submitted 2017-11-14; First posted 2018-05-16 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Cognitive Function; Mood
Keywords: Cognition; Mood; Flavonoid; Grape Seed; Catechin; Epicatechin; Proanthocyanidin

STUDY DESIGN:
Intervention Model Description: Acute on chronic
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CP9700 (Experimental): 400 mg CP9700 along with modified cellulose (MCC), magnesium stearate, silica (sillicon dioxide), Gelatin, FD&C Red No. 40, titanium dioxide, sodium lauryl sulfate, glycerin, brilliant blue FCF consumed with breakfast in a 1 capsule per day regimen.
  Interventions: Dietary Supplement: CP9700
- Matched Placebo (Placebo Comparator): Maltodextrin along with modified cellulose (MCC), magnesium stearate, silica (sillicon dioxide), Gelatin, FD&C Red No. 40, titanium dioxide, sodium lauryl sulfate, glycerin, brilliant blue FCF consumed with breakfast in a 1 capsule per day regimen.
  Interventions: Dietary Supplement: Matched Placebo

INTERVENTIONS:
Dietary Supplement: CP9700 — 400 mg CP9700 along with modified cellulose (MCC), magnesioum strearate, slica (sillicon dioxide), Gelatin, FD&C Red No. 40, titanium dioxide, sodium lauryl sulfate, glycerin, brilliant blue FCF consumed with breakfast in a 1 capsule per day regimen.
  Arms: CP9700
Dietary Supplement: Matched Placebo — Maltodextrin along with modified cellulose (MCC), magnesioum strearate, slica (sillicon dioxide), Gelatin, FD&C Red No. 40, titanium dioxide, sodium lauryl sulfate, glycerin, brilliant blue FCF consumed with breakfast in a 1 capsule per day regimen.
  Arms: Matched Placebo

SUMMARY:
This acute-on-chronic study will examine the effectiveness of CP9700 for improving cognitive performance and mood in healthy young adults. CP9700 is a mix of highly purified grape seed-derived polyphenolic extracts from Vitis vinifera produced by Polyphenolics Inc. (Madera, CA, USA). The polyphenolic component of the product is comprised entirely of catechin and epicatechin, derivatives of catechin and epicatechin (e.g.,epicatechin gallate), and proanthocyanidins. We will perform a randomised, double-blind, parallel-groups human intervention trial using CP9700 and a well characterised sugar-matched placebo to investigate changes in cognitive performance.

DETAILED DESCRIPTION:
Interventions: Two interventions will be tested, CP9700 (400 mg) and a placebo. Importantly, the placebo will be matched to the active treatment for sugars and vitamin C levels. All interventions will be supplied in blister packs.

Participants: A total of 60 healthy, young adult participants will be recruited for these studies. Based upon the medium effect size (d = .65) observed in previous work using healthy adults and the Go/No go task, we calculate that a sample of 25 participants/treatment will provide considerable power (.70) to detect a similar sized effect in this study. The recruitment procedure allows for a 15% drop out rate. Participants will be recruited directly from the School of Psychology & Clinical Language Sciences Undergraduate Research Panel.

Procedure: Following recruitment to the study, participants will start a two-week 'run-in' phase. During this phase, all participants will complete a 3-day food frequency questionnaire to give a measure of their habitual diet before being asked to adhere to a low-flavonoid diet, we will collect a 3-day food diary to check compliance and they will attend the laboratory for an initial 'practice' session of the cognitive tasks (see below). On the evening before the 'active treatment' phase commences, participants will be asked to consume a standard meal- this procedure will be repeated for each evening meal consumed prior to a test day. On the acute test day, participants will attend the laboratory in a fasted state where they will receive a standard low-flavanoid breakfast, followed by a battery of cognitive and mood tasks (see below). Subjects will then be given their intervention, and will be re-tested on our task battery at two-hourly intervals over a 6 hour period before being allowed to return home. During the chronic phase of the study, after 6 and 12 weeks of consuming the intervention, subjects will return to the lab in a fasted state (prior to taking their daily intervention), will be given a standard low flavonoid breakfast, and will be tested on the task battery before consuming their allocated intervention. Compliance will be assured through collection of used blister packs.

The task battery is composed of cognitive tests and measures of mood, which our previous data show to be sensitive to flavonoid interventions, both acutely and chronically. More generally, the cognitive tests are categorised into one of two key cognitive domains; (i) Executive Function (i.e., Serial Sevens, Stroop, Modified Attention Network Test) and (ii) Episodic Memory (i.e., immediate and delayed auditory recall, verbal recognition, immediate and delayed spatial memory). Moreover, our previous data indicates increased cerebral blood flow in the in the acute postprandial phase 2-5 hours following flavonoid consumption in brain regions required for executive function and episodic memory including the frontal cortex and frontal gyrus. In addition, changes in mood will be measured using the PANAS, which has previously been shown to be sensitive to flavonoid interventions acutely and chronically.

ELIGIBILITY:
Inclusion Criteria:

* Non Smoker
* Not Pregnant
* Non vegetarian or vegan
* Able to consume the capsules

Exclusion Criteria:

* Should not suffer from any of the following diseases: Major mental illness; Liver disease; Diabetes mellitus (Type 1 and 2); Heart disease; Renal or gastrointestinal disorders
* Should not be taking blood pressure lowering or anticoagulant medication
* Should not be taking depression medication
* Should not be consuming more than the Government recommended units of alcohol per week
* Should not be vigorous exercisers (restricted to < 4 hours per week for the duration of the study)
* Should not be taking nutritional supplements (for the duration of the study)
* Should not be taking recreational drugs (either illegal or legal for the duration of the study)

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Cognitive Performance - Episodic Memory | 2 hrs following acute intervention.
  As Measured by the Auditory Verbal Learning Task
Cognitive Performance - Episodic Memory | 4 hrs following acute intervention.
  As Measured by the Auditory Verbal Learning Task
Cognitive Performance - Episodic Memory | 6 hrs following acute intervention.
  As Measured by the Auditory Verbal Learning Task
Cognitive Performance - Episodic Memory | Following 6 weeks chronic intervention
  As Measured by the Auditory Verbal Learning Task
Cognitive Performance - Episodic Memory | Following 12 weeks chronic intervention
  As Measured by the Auditory Verbal Learning Task
Cognitive Performance - Attention shifting | 2 hrs following acute intervention.
  As measured by the Switching Task
Cognitive Performance - Attention shifting | 4 hrs following acute intervention.
  As measured by the Switching Task
Cognitive Performance - Attention shifting | 6 hrs following acute intervention.
  As measured by the Switching Task
Cognitive Performance - Attention shifting | Following 6 weeks chronic intervention
  As measured by the Switching Task
Cognitive Performance - Attention shifting | Following 12 weeks chronic intervention
  As measured by the Switching Task
Cognitive Performance - Motor Control | 2 hrs following acute intervention.
  As measured by the finger tapping task
Cognitive Performance - Motor Control | 4 hrs following acute intervention.
  As measured by the finger tapping task
Cognitive Performance - Motor Control | 6 hrs following acute intervention.
  As measured by the finger tapping task
Cognitive Performance - Motor Control | Following 6 weeks chronic intervention
  As measured by the finger tapping task
Cognitive Performance - Motor Control | Following 12 weeks chronic intervention
  As measured by the finger tapping task
Cognitive Performance - Working Memory | 2 hrs following acute intervention.
  As measured by the serial 3 and 7s task
Cognitive Performance - Working Memory | 4 hrs following acute intervention.
  As measured by the serial 3 and 7s task
Cognitive Performance - Working Memory | 6 hrs following acute intervention.
  As measured by the serial 3 and 7s task
Cognitive Performance - Working Memory | Following 6 weeks chronic intervention
  As measured by the serial 3 and 7s task
Cognitive Performance - Working Memory | Following 12 weeks chronic intervention
  As measured by the serial 3 and 7s task
Cognitive Performance - Visual Memory Span | 2 hrs following acute intervention.
  As measured by the Corsi Block Task
Cognitive Performance - Visual Memory Span | 4 hrs following acute intervention.
  As measured by the Corsi Block Task
Cognitive Performance - Visual Memory Span | 6 hrs following acute intervention.
  As measured by the Corsi Block Task
Cognitive Performance - Visual Memory Span | Following 6 weeks chronic intervention
  As measured by the Corsi Block Task
Cognitive Performance - Visual Memory Span | Following 12 weeks chronic intervention
  As measured by the Corsi Block Task

SECONDARY OUTCOMES:
Mood | 2 hrs following acute intervention.
  As measured by the Positive and Negative Affect Schedule
Mood | 4 hrs following acute intervention.
  As measured by the Positive and Negative Affect Schedule
Mood | 6 hrs following acute intervention.
  As measured by the Positive and Negative Affect Schedule
Mood | Following 6 weeks chronic intervention
  As measured by the Positive and Negative Affect Schedule
Mood | Following 12 weeks chronic intervention
  As measured by the Positive and Negative Affect Schedule

CONTACTS AND LOCATIONS:
Overall Officials: Claire M Williams, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macready AL, Kennedy OB, Ellis JA, Williams CM, Spencer JP, Butler LT. Flavonoids and cognitive function: a review of human randomized controlled trial studies and recommendations for future studies. Genes Nutr. 2009 Dec;4(4):227-42. doi: 10.1007/s12263-009-0135-4. Epub 2009 Aug 13. PMID 19680703
- [Background] Bell L, Lamport DJ, Butler LT, Williams CM. A Review of the Cognitive Effects Observed in Humans Following Acute Supplementation with Flavonoids, and Their Associated Mechanisms of Action. Nutrients. 2015 Dec 9;7(12):10290-306. doi: 10.3390/nu7125538. PMID 26690214
- [Background] Lamport DJ, Dye L, Wightman JD, Lawton CL. A. The effects of flavonoid and other polyphenol consumption on cognitive performance: A systematic research review of human experimental and epidemiological studies. Nutrition and Aging. 1(1), 5-25, 2012